CLINICAL TRIAL: NCT00218348
Title: Pharmacotherapy for Cocaine Dependence - 1
Brief Title: Treatment of Cocaine Dependence: Comparison of Three Doses of Dextro-Amphetamine Sulfate and Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joy Schmitz, Professor - Psy, Behavioral Science, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-16305-1; R01DA016305 (NIH); R01-16305-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Abuse; Dextro-Amphetamine Sulfate
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Dextroamphetamine

INTERVENTIONS:
Drug: Dextro-Amphetamine Sulfate

SUMMARY:
Dextro-amphetamine sulfate is a central nervous system stimulant that increases the release of the neurotransmitter dopamine in the brain. The purpose of this study is to further examine dose ranges of dextro-amphetamine sulfate as a treatment for cocaine dependence.

DETAILED DESCRIPTION:
This randomized, double-blind dose study will compare the effectiveness of three active medication doses of dextro-amphetamine sulfate to placebo in the treatment of cocaine dependence. Participants will be randomly assigned to one of the four following dosages of dextro-amphetamine sulfate: 0 mg, 40 mg, 60 mg, or 80 mg. Participants will undergo a 2-week stabilization period followed by a 25-week study period. The study period will include administration of the stable medication dose for 21 weeks, followed by 1 week of dose reduction, and then 3 weeks without medication. All participants will receive weekly cognitive behavioral therapy and electrocardiograms. Participants will be given the option to participate in a voluntary plasma blood draw during Weeks 4, 8, and 20 and will be scheduled for follow-up assessments at Months 1 and 3 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of cocaine dependence, as determined by the Structured Clinical Interview for DSM-IV
* Agreement to use an adequate method of contraception for the duration of the study
* Electrocardiogram confirmation by a cardiologist
* Cocaine-positive urine test prior to study entry

Exclusion Criteria:

* High blood pressure
* Significant heart disease
* Clinically significant cardiovascular abnormality
* Angina
* Kidney, liver, or gastrointestinal disorder
* Current Axis I disorder not related to drug use
* Current dependence on any drug other than nicotine
* Attention deficit disorder (ADD) or attention deficit hyperactivity disorder (ADHD)
* On probation or parole for reasons other than those related to drug abuse charges
* Pregnant or breastfeeding
* Sought treatment for drug dependence within 3 months prior to study entry
* Currently taking prescribed medications

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2003-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Substance use and retention

SECONDARY OUTCOMES:
Effectiveness measures, including psycho-social variables, side effects, and self-reported measures

CONTACTS AND LOCATIONS:
Overall Officials: Joy M Schmitz, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States